CLINICAL TRIAL: NCT04067167
Title: Effects of Flexi Band Resistance Training Versus Different Electromyostimulation Exercise Programs in Patients With the Diagnosis of Malignant Diseases
Brief Title: Flexi Band Resistance Training Versus EMS Exercise in Patients With the Diagnosis of Malignant Diseases
Acronym: FREEDOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FREEDOM-Study
Record Dates: First submitted 2019-05-15; First posted 2019-08-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Cancer Cachexia; Inflammation; Muscular Atrophy
Keywords: Cancer; Cachexia; Muscular strength; Resistance training; Body composition; Muscle mass; Physical exercise; Nutrition; whole-body electromyostimulation
MeSH Terms: conditions — Neoplasms; Inflammation; Muscular Atrophy; Cachexia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment parallel-group, randomized-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WB-EMS (Sham-intervention) (Sham Comparator): Low-theshold WB-EMS combined with nutritional therapy
  Interventions: Other: WB-EMS (Sham-intervention)
- WB-EMS (Experimental): WB-EMS combined with nutritional therapy
  Interventions: Other: WB-EMS
- Free WB-EMS (Experimental): WB-EMS using a mobile System combined with nutritional therapy
  Interventions: Other: Free WB-EMS
- Flexi Band Resistance Training (Experimental): Flexi band resistance Training combined with nutritional therapy
  Interventions: Other: Flexi band resistance training

INTERVENTIONS:
Other: WB-EMS (Sham-intervention) — Whole-Body Electromyostimulation (WB-EMS):
  WB-EMS with low-threshold stimulation during a study period of 12 weeks combined with standard nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted Protein intake/day: 1.2 - 1.5 g per kg bodyweight)
  * patients perform simple exercises during the stimulation period following a video tutorial
  * time-effort per session: ~20 min
  * 2 training sessions per week
  Arms: WB-EMS (Sham-intervention)
Other: WB-EMS — Whole-Body Electromyostimulation (WB-EMS):
  WB-EMS during study period of 12 weeks combined with standard nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted Protein intake/day: 1.2 - 1.5 g per kg bodyweight)
  * WB-EMS stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec;
  * patients perform simple exercises during the stimulation period following a video tutorial
  * time-effort per session: ~20 min
  * 2 training sessions per week
  Arms: WB-EMS
Other: Free WB-EMS — Whole-Body Electromyostimulation (WB-EMS) using a mobile system:
  WB-EMS during study period of 12 weeks combined with standard nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted Protein intake/day: 1.2 - 1.5 g per kg bodyweight)
  * WB-EMS stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec;
  * patients perform simple exercises during the stimulation period following a video tutorial
  * time-effort per session: ~20 min
  * 2 training sessions per week
  Arms: Free WB-EMS
Other: Flexi band resistance training — Flexi band resistance Training:
  Training during study period of 12 weeks combined with standard nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted Protein intake/day: 1.2 - 1.5 g per kg bodyweight)
  * patients perform resistance exercises using flexi bands
  * flexi band exercises are conceptualized to activate similar muscle groups as EMS exercise
  * time-effort per session: ~20 min
  * 2 training sessions per week
  Arms: Flexi Band Resistance Training

SUMMARY:
The purpose of this study is to investigate the effects of a 12-week flexi band resistance training program compared to different whole-body electromyostimulation (WB-EMS) exercise programs on muscle strength, body composition (in particular muscle mass), cardiorespiratory fitness, inflammation, and patient-reported subjective outcomes (e.g. quality of life, fatigue, performance status) in patients with malignant disease undergoing curative or palliative anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* malignant disease (solid or hematological cancer): head and neck cancer, colorectal carcinoma, small intestinal cancer, gastric cancer, oesophageal cancer, pancreas carcinoma, liver cell carcinoma, cholangiocarcinoma, lung cancer, breast cancer, cervix cancer, ovarian cancer, prostate cancer, renal cell carcinoma, malignant melanoma, patients with leukaemia and malignant lymphomas or Graft-versus-Host-Disease after bone marrow transplantation
* ongoing or planned curative or palliative anti-cancer therapy
* ECOG-Status 0-2

Exclusion Criteria:

* simultaneous participation in other nutritional or exercise intervention Trials
* bone metastases with high fracture risk
* cardiovascular disease
* use of anabolic medications
* epilepsy
* severe neurological or rheumatic diseases
* skin lesions in the area of electrodes
* energy active metals in body
* pregnancy
* acute vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 12 weeks
  Muscle strength of the five major muscle groups (chest, upper back, lower back, abdominals, legs) will be assessed by using specific strength-training devices and estimated using the one Repetition Maximum (1-RM, the maximum amount of weight [kg] that can be lifted for one repetition)

SECONDARY OUTCOMES:
Muscle Mass | 12 weeks
  Muscle mass (kg) will be measured by Bioelectrical Impedance Analysis (BIA)
Fat Mass | 12 weeks
  Fat mass (kg) will be measured by Bioelectrical Impedance Analysis (BIA)
Total Body Water | 12 weeks
  Total body water (L) will be measured by Bioelectrical Impedance Analysis (BIA)
Cardiorespiratory Fitness (CRF) | 12 weeks
  CRF will be assessed by measuring Maximum Oxygen uptake (VO2max)
Inflammation status | 12 weeks
  Inflammation will be assessed by measuring blood levels (mg/L) of c-reactive protein (CRP) and high-sensitivity c-reactive protein (hs-CRP).
Patient-reported performance status-1 | 12 weeks
  Patient-reported performance Status will be assessed using the ECOG Performance Status questionnaire. It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. The score ranges from 0-5 (lower values = better outcome).
Patient-reported performance status-2 | 12 weeks
  Patient-reported performance status-2 will be assessed using the Karnofsky index. It is used methods to assess the functional status of a Patient. The score ranges from 0-100 (higher value = better outcome).
Patient-reported Quality of Life (QoL) | 12 weeks
  Patient-reported QoL will be assessed using the EORTC QLQ-C30 questionnaire. It contains 30 questions (items), representing various aspects/dimensions of QoL (physical, role, emotional, cognitive and social), and 3 symptom scales (fatigue, pain and nausea).The scales of the different dimensions of QoL (higher values = better outcome) and symptoms (lower values = better outcomes) range from 0-100.
Patient-reported Fatigue | 12 weeks
  Fatigue will be assessed using the FACIT-Fatigue scale. It contains 13 items (different aspects/dimensions of fatigue) each assessed on a scale of 0-4, with lower values indicating a better outcome).
Patient-reported Physical Activity | 12 weeks
  Patient-reported Physical Activity (PA) will be assessed using the the International Physical Activity Questionnaire (IPAQ). IPAQ records 4 aspects of PA (job-, transportation-, housework-, and leisure-time-related). There are two forms of output from scoring the IPAQ. Results can be reported in categories (low, moderate or high PA levels) or as a continuous variable (MET minutes a week, 1 MET = resting energy expenditure). MET minutes represent the amount of energy expended carrying out physical activity. High PA = at least 1500 MET minutes/week; moderate PA: at least 600 MET minutes/week; low PA: < 600 MET minutes/week. Higher values represent a better outcome.
Objective Physical Activity | 12 weeks
  Obejective measurement of physical activity will be preformed using Pedometers. Higher values represent a better outcome.
Cardiometabolic Risk Profile (Metabolic Syndrome Z-Score, MetS) | 12 weeks
  MetS will be calculated MetS-Z-Score will be calculated from each individual's measures of waist circumference (cm), mean arterial blood pressure (mmHg), blood levels of glucose (mg/dL), triglycerides (mg/dL), and HDL-cholesterol (mg/dL), based on equations specific to sex.

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Reljic, Dr., Principal Investigator — University Erlangen Nuremberg Medical School; Yurdagül Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector-Center for Nutrition, Exercise and Sports, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939